CLINICAL TRIAL: NCT05431998
Title: Evaluation of Autogenous Demineralized Tooth Graft Versus Autogenous Bone Graft During Immediate Implant Placement in the Esthetic Zone. (Randomized Controlled Clinical Trial).
Brief Title: Evaluation of Autogenous Demineralized Tooth Graft Versus Autogenous Bone Graft During Immediate Implant Placement in the Esthetic Zone.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Taha Taha Ahmed, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: At1
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Estetic Zone; Autogenous Tooth Graft; Autogenous Bone Graft; Immediate Implant; Jumping Gap; Crestal Bone Level

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The use of demineralized autogenous tooth graft in the jumping gap of the immediate implant (Experimental): The participant's own freshly extracted tooth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries, or restorations (if present) and have their crown decapitated, using a high-speed fine finishing stone and saline irrigation. The pulp chamber and root pulp will be cleaned by split opening the root and cleaning it out using a high-speed diamond bur. Subsequently, teeth will be ground, and demineralized using a hand bone mill (Gold Bone Mill, MCT Bio, Korea). Then the particles will be prepared by demineralization of tooth particles in 0.6N hydrochloric acid (Chemajet Chemicals, Egypt) for 30 min then washed twice in saline and dried with sterile gauze. Then it will be used as a graft for the bone defect around the immediately placed implant.
  Interventions: Procedure: the use of demineralized autogenous tooth graft in the jumping gap during immediate implant placement
- The use of autogenous bone graft in the jumping gap of the immediate implant (Active Comparator): A horizontal vestibular incision will be placed below the mucogingival junction and a mucoperiosteal flap will be reflected then autogenous bone particles will be collected from the participants using Automatic Bone Collector Bur (ACM Bur) by NeoBiotch, from the mandibular retro-molar region, speed 300rpm, torque 30Ncm, with irrigation.
  Interventions: Procedure: the use of autogenous bone graft in the jumping gap during immediate implant placement

INTERVENTIONS:
Procedure: the use of demineralized autogenous tooth graft in the jumping gap during immediate implant placement — the use of demineralized autogenous tooth graft in the jumping gap during immediate implant placement
  Arms: The use of demineralized autogenous tooth graft in the jumping gap of the immediate implant
Procedure: the use of autogenous bone graft in the jumping gap during immediate implant placement — the use of autogenous bone graft in the jumping gap during immediate implant placement
  Arms: The use of autogenous bone graft in the jumping gap of the immediate implant

SUMMARY:
To compare the use of demineralized autogenous tooth graft versus autogenous bone graft, in the jumping gap in immediate implant placement with immediate loading.

DETAILED DESCRIPTION:
Immediate implant placement was introduced in 1978, using a ceramic implant made of Al2O3. Ever since then it has become one of the most successful treatment options to maintain the alveolar bone after tooth extraction, showing success rate of more than 95%. Continuous research and development of immediate implant techniques keep being introduced, stemming from the fact that immediate implant placement is a safe, predictable, and favorable solution after the loss of a tooth.

A 2 mm jumping gap is recommended in the treatment guidelines proposed in an ITI Consensus Conference. This provides sufficient space to fill the bone defect between the exposed implant surface and the facial bone wall with an appropriate bone filler. A gap in these dimensions also provides a space for the formation of a blood clot which can subsequently reorganize into a provisional connective tissue matrix and support the formation of newly formed woven bone. This was demonstrated in a preclinical study in which a wider defect and bone wall dimension were associated with less crestal bone height reduction and more bone to implant contact than a narrower defect and bone wall dimension. Also, immediate placement with a dual-zone augmentation technique, and a socket seal technique utilizing a prefabricated shell made of acrylic and immediate restoration, out of occlusion showed very promising results.

The addition of graft material during immediate implant placement is very common and useful in many cases. Autogenous bone graft is considered to be the gold standard graft material, which makes comparing new graft materials to it sensible. Still, tooth bone graft has been used numerous of times for socket preservation, and it shows good results.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of extraction of a single, un-restorable tooth in the esthetic zone (Maxillary anteriors and premolars). Only one implant per patient.

An intact buccal plate of bone, or minimally affected. Jumping gap ≥ 2mm . Age 18-60. Medically free patients.

Exclusion Criteria:

* Restorable teeth. Teeth with severely damaged or no remaining buccal plate. Acute infection in the implant site. Patients with an insufficient bone to obtain primary stability. Patients in need of sinus bone grafting. A systemic condition that affects bone healing (e.g., diabetes mellitus or bone disease).

Smokers. Poor oral hygiene. Patient with a physical disability that hinders the upkeep of good oral hygiene measures.

Any general contraindication to oral surgery. Participants suffering from diseases that may affect bone or soft tissue healing.

A participant who had radiotherapy or chemotherapy. Psychiatric patient, or with a learning disability, or unable to give consent. Pregnant and nursing women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level | 9 months
  Marginal bone level: The bone level will be measured from the implant shoulder to the first bone-implant contact, from all 4 surfaces (mesial, distal, buccal, and lingual/palatal), measured by CBCT scans.

SECONDARY OUTCOMES:
post operative pain | 2 weeks
  Visual analog scale (0-10)
Implant sucess | 12 months
  Based on the criteria of Albrektsson, Zarb, Worthington, and Eriksson(1986) and of Buser, Weber and Lang(1990). The following are the criteria for implant success: the absence of mobility, the absence of acute or chronic peri-implant infection, the absence of radiolucency around the implant, without pocket probing depth (PPD) ≧ 5 mm, and without vertical bone loss ≧ 1.5 mm in the first year. The cases will be defined as a failure if they can't reach any one of the success criteria
Pink esthetic score | 12 months
  The PES includes seven variables: the mesial papilla, distal papilla, midfacial level, midfacial contour, alveolar process deficiency, soft tissue color, and soft tissue texture. Each variable was evaluated with a 0-1-2 score, with 2 being the best and 0 being the worst. Thus, the highest total score was 14. The mesial and distal papillae were assessed for completeness. All other variables were evaluated by comparison with the contralateral tooth. The threshold of an acceptable PES was 8. Scores of 12 or more indicated a nearly perfect outcome

CONTACTS AND LOCATIONS:
Overall Officials: Karim M Fawzy, PhD, Study Chair — Cairo University; Nesma M Shemais, PhD, Study Director — Cairo University; Rahma H Ahmed, BDS, Principal Investigator — Cairo University; Ahmed T Taha, BDS, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry Ciaro University, Cairo, El Manial, Egypt